CLINICAL TRIAL: NCT02110680
Title: Efficacy of Transcutaneous Nerve Stimulation on Improvement of Overactive Bladder Symptoms
Acronym: TENSOAB
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, MICHAEL VAINRIB, M.D., Meir Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: TENSOAB; TENSOAB (Other: 0228-13MMC)
Record Dates: First submitted 2014-03-28; First posted 2014-04-10 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; transcutaneous electric stimulation; posterior tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- TENS 1 (Active Comparator): TENS at posterior tibial nerve area
  Interventions: Device: Sports TENS 2
- TENS 2 (Sham Comparator): TENS at shoulder area
  Interventions: Device: Sports TENS 2

INTERVENTIONS:
Device: Sports TENS 2 — transcutaneous electric stimulation
  Other Names: Sports TENS 2 by TensCare Ltd, United Kingdom.

SUMMARY:
Overactive bladder (OAB) is a very common problem that impairs the quality of life of about 17% of adult population in USA above the age of 40. The issues becomes more prominent with getting older. OAB was determined by International Continence Society as urgency (immediate desire to urinate that could not be postponed) with or without incontinence usually associated with increased frequency and nocturia (urination at night). In 2012, American Urologic Association published clinical guidelines for the treatment of OAB of non neurogenic origin. Neuromodulation was proposed as the third line of treatment and two treatments were recommended: sacral nerve neuromodulation (SNM) and posterior tibial nerve stimulation (PTNS). Each of above mentioned procedures are invasive. SNM involves lead implantation in operating room using X-ray guidance and anesthesia. PTNS involves needle insertion on the low extremity.

The investigators would like to examine the efficacy of transcutaneous nerve stimulation (TENS) in refractory to the first two lines of OAB treatment patients.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients
* age above 18
* OAB symptoms more than 6 months before run into the study
* OAB symptoms refractory to medical oral and cognitive treatments
* Adverse events or unwillingness to continue with abovementioned treatments
* patients with OAB symptoms with no evidence of neuropathic nature
* patients who signed informed consent fully understanding the treatment and study design

Exclusion Criteria:

* children
* patients who unable or did not sign an informed consent or do not understand the study design and the treatment
* patients who have implanted electric devices (eg. cardiac stimulators etc.)
* patients who have post voiding residual more than 100ml
* patients who have neuropathic OAB or pelvic ongoing malignancy or prior pelvic radiation
* patients who were treated in the last 6 months with SNM, PTNS or intravesical Botox injections
* patients with denovo OAB after recent implantation of tension-free vaginal tape (TVT) procedure
* stress urinary incontinence predominant complaints in mixed incontinence patients
* significant pelvic organ prolapse in women or an evidence of significant bladder outlet obstruction in male patients
* patients with a history of recurrent urinary tract infections (UTIs) during the last 2 years
* any medical condition that involves skin on the lower extremity
* bilateral leg amputation
* any medical condition that on investigator's mind could have an adverse impact on the patient during the study
* participation in a clinical study at the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in day and night-time frequency of micturitions | 12 weeks
  change in OAB-q (overactive bladder questionnaire) score bladder diary: change in a frequency of micturitions during the day and night. change in a mean volume of micturitions.
Change in a number of urgency and urge incontinence episodes | 12 weeks
  change in OAB-q (overactive bladder questionnaire) score bladder diary: change in a number of urgency and urge incontinence episodes

SECONDARY OUTCOMES:
Change in quality of life in patients with overactive bladder syndrome at the end of TENS treatment | 12 weeks
  Filling of questionnaires: OAB-q (overactive bladder questionnaire), Patient perception of bladder condition (PPBC), Patient perception of global improvement (PPGI), Quality of life 5 dimensions (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vainrib, M.D., Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel